CLINICAL TRIAL: NCT01362348
Title: An Open-label, Phase 2a Study to Evaluate Pazopanib Eye Drops Administered for 12 Weeks to Patients With Neovascular Age-related Macular Degeneration
Brief Title: 12 Week Patient Study in Neovascular Age-related Macular Degeneration (AMD)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Lack of efficacy identified during a preliminary analysis
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 114987
Record Dates: First submitted 2011-05-19; First posted 2011-05-30 (Estimated); Results first posted 2017-08-21 (Actual); Last update posted 2017-09-21 (Actual); Status verified 2017-08

CONDITIONS: Macular Degeneration
Keywords: Age-related Macular Degeneration
MeSH Terms: conditions — Macular Degeneration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- pazopanib eye drops (Experimental): pazopanib topical ocular administration
  Interventions: Drug: pazopanib eye drops

INTERVENTIONS:
Drug: pazopanib eye drops — 10 mg/mL (1 drop) four times daily

SUMMARY:
The purpose of this 12 week, open-label study is to investigate the safety and efficacy of a single dose regimen of pazopanib eye drop for neovascular AMD.

DETAILED DESCRIPTION:
MD7114987 is a Phase 2a study designed to determine whether pazopanib eye drops have the potential to reduce retinal edema and maintain or improve visual acuity in persons with a previously untreated subfoveal choroidal neovascularization (CNV) lesion secondary to age-related macular degeneration (AMD) and to further characterize the safety and tolerability of pazopanib eye drops administered over a 12-week period.

ELIGIBILITY:
Inclusion Criteria:

Subjects eligible for enrolment in the study must meet all of the following criteria:

* Consent: Subject understands the procedures, agrees to participate in the study (including participation in the CFH Y402H pharmacogenetic research), and has signed and dated the informed consent form prior to the initiation of any study-related activities. If the subject is unable to read the consent form due to visual impairment then the consent must be read to the subject verbatim by the person administering the consent, a family member, or legally acceptable representative. (Note: Consent by legally acceptable representative is allowed where this is in accordance with local laws, regulations, and ethics committee policy.)
* Age-related macular degeneration: For each subject enrolled in the study, only one eye (study eye) will be treated, and eligibility criteria apply to the study eye. All of the following characteristics are required and must be confirmed by the central reading center:
* CNV caused by AMD that extends under the geometric center of the foveal avascular zone
* Center subfield thickness (inclusive of subretinal fluid) > 320 microns on OCT [SPECTRALIS® (Heidelberg)]
* Total lesion area ≤12 disc areas on fluorescein angiography, where the lesion complex includes CNV, blood, blocked florescence not from blood, and serous detachment of the retinal pigment epithelium
* CNV comprises < 50% of lesion area
* classic CNV comprises < 50% of the lesion area
* fibrosis comprises ≤ 25% of lesion area
* if no evidence of classic CNV, then presumed to have recent disease progression based on deterioration (≥ 5 letter decrease in vision or evidence of growth of a CNV lesion on fluorescein angiography ) within the last 3 months or evidence of hemorrhage from CNV
* Visual acuity: Best-corrected visual acuity score by electronic ETDRS in the study eye of between 25 and 73 letters (approximately equivalent to Snellen VA of 20/320 to 20/32) at screening
* Gender and age: Subject is a male or female adult 50 years of age or older.
* Non-childbearing potential: Female subject is of non-childbearing potential defined as being physiologically incapable of becoming pregnant. This includes any female who is post-menopausal (12 months of spontaneous amenorrhea) or who is surgically post-menopausal (via documented hysterectomy or bilateral tubal ligation). In questionable cases of postmenopausal status, a blood sample with simultaneous follicle stimulating hormone (FSH) >40 MIU/mL and estradiol <40 pg/mL (<140 pmol/L) [or equivalent values based on local laboratory criteria] is confirmatory. Refer to the SPM for more information.
* Study Compliance: Subject is able and willing to comply with the study requirements and is able and willing to attend all scheduled visits.
* Liver function tests: Subject has liver chemistry values that are within normal limits or clinically insignificant as evidenced by serum aspartate aminotransferase (AST) and alanine aminotransferase (ALT) <2xULN; alkaline phosphatase and bilirubin <1.5xULN (isolated bilirubin >1.5xULN is acceptable, if bilirubin is fractionated and direct bilirubin is < 35%).
* QT interval: Subject has a QTcF value < 450 msec, or < 480 msec for subjects with Bundle Branch Block. [Note: subjects with paced rhythms may be considered pending discussion with the medical monitor.]

Exclusion Criteria:

Subjects meeting any of the following criteria must not be enrolled in the study:

Study Eye:

* Additional eye disease in the study eye that could compromise best-corrected visual acuity (e.g. glaucoma with documented visual field loss, clinically significant diabetic retinopathy, ischemic optic neuropathy, infection or retinitis pigmentosa)
* CNV in the study eye due to other causes unrelated to age-related macular degeneration
* Presence of retinal angiomatous proliferation (RAP) in the study eye, as determined by the investigator (confirmation by indocyanine green angiography is not required)
* Geographic atrophy involving the center of the fovea in the study eye
* Anterior segment and vitreous abnormalities in the study eye that would preclude adequate observation of the fundus for photographs, fluorescein angiography and spectral-domain OCT
* Vitreous, subretinal or retinal hemorrhage in the study eye that is unrelated to AMD
* Presence of an RPE tear in the study eye
* Aphakia or total absence of the posterior capsule (Yttrium aluminum garnet (YAG) capsulotomy permitted) in the study eye
* History of vitrectomy in the study eye
* Intraocular surgery in the study eye within 3 months prior to treatment
* Any previous treatment in the study eye for neovascular AMD, approved or investigational

Fellow Eye:

* Current intravitreal anti-VEGF therapy in the fellow eye
* Best-corrected visual acuity score by electronic ETDRS < 56 letters in the fellow eye at screening

Concurrent Conditions or Concomitant Medications:

* Subject has uncontrolled glaucoma (intraocular pressure > 25 mmHg) despite treatment with anti-glaucoma medication.
* A known, positive test for Hepatitis B surface antigen or Hepatitis C antibody within 3 months of screening
* Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones)
* Active bleeding disorder or a history of hemoptysis, cerebral or clinically significant gastrointestinal hemorrhage within 6 months of screening
* Significant uncontrolled or unstable cardiovascular, nervous system, pulmonary, renal, endocrine, or gastrointestinal disease for example:
* Uncontrolled diabetes mellitus, with hemoglobin A1c (HbA1c) > 10%
* Myocardial infarction or stroke within 6 months of screening
* Major surgery within 3 months of screening
* Clinically relevant thyroid disease
* Uncontrolled hypertension:

Systolic blood pressure > 160 mmHg Diastolic blood pressure > 100 mmHg Note: Initiation or adjustment of antihypertensive medications is permitted prior to study entry provided the referenced criteria are met (See Section 4.4.3).

* Subject has a history within the past 2 years of alcohol or substance abuse, or psychiatric disorder likely to confound the efficacy or safety assessments.
* Known HIV infection
* Within 6 months prior to the Screening Visit, use of any systemically administered anti angiogenic agent (e.g., bevacizumab, sunitinib, cetuximab, sorafenib, pazopanib), approved or investigational
* Within 6 months prior to the Screening Visit, use of medications known to be toxic to the retina, lens or optic nerve (e.g. desferoximine, chloroquine/hydrochloroquine, chlorpromazine, phenothiazines, tamoxifen, and ethambutol)
* Use of systemic steroids (>10 mg prednisone or equivalent/day) within 14 days of the start of treatment
* Use of prohibited medications within the restricted timeframe relative to the start of study medication (See Section 5.5.2)
* Use of an investigational drug within 30 days of screening
* History of sensitivity to any of the study medications, or components thereof or a history of drug or other allergy that, in the opinion of the investigator or GSK Medical Monitor, contraindicates their participation
* A condition or situation, which, in the opinion of the investigator, may result in significant risk to the patient, confound the study results or interfere significantly with participation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-07-07 (Actual); Primary Completion 2012-04-16 (Actual); Study Completion 2012-04-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (14):
- United States (9):
  - GSK Investigational Site, Phoenix, Arizona
  - GSK Investigational Site, Miami, Florida
  - GSK Investigational Site, Winter Haven, Florida
  - GSK Investigational Site, Decatur, Georgia
  - GSK Investigational Site, Boston, Massachusetts
  - GSK Investigational Site, Grand Rapids, Michigan
  - GSK Investigational Site, Cleveland, Ohio
  - GSK Investigational Site, Austin, Texas
  - GSK Investigational Site, Houston, Texas
- GSK Investigational Site, Paris, France
- Germany (4):
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Münster, North Rhine-Westphalia
  - GSK Investigational Site, Leipzig, Saxony

REFERENCES:
- [Derived] Singh R, Wurzelmann JI, Ye L, Henderson L, Hossain M, Trivedi T, Kelly DS. Clinical evaluation of pazopanib eye drops in healthy subjects and in subjects with neovascular age-related macular degeneration. Retina. 2014 Sep;34(9):1787-95. doi: 10.1097/IAE.0000000000000179. PMID 24896137

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study was conducted at 10 sites in the United States, Germany and France from 7 July 2011 was early terminated on 22 Mar 2012 and completed on 16 April 2012. The study was terminated due to lack of efficacy.
Groups:
- Pazopanib 10 mg/mL QID: Eligible participants instilled a single drop (approximately 40 micro liters ) of the pazopanib ophthalmic solution 10 milligram per millimeter (mg/mL) via topical ocular route to the study eye at approximate 5 hour intervals four times a day (QID) during the non-sleep period for a duration of 12 weeks.
Period: Overall Study
Arm/Group | Pazopanib 10 mg/mL QID
Started | 19
Completed | 5
Not Completed | 14
Not completed — Protocol-defined stopping criteria | 9
Not completed — Study closed/terminated | 5

BASELINE CHARACTERISTICS:
Groups:
- Pazopanib 10 mg/mL QID: Eligible participants instilled a single drop (approximately 40 microliters ) of the pazopanib ophthalmic solution 10 mg/mL via topical ocular route to the study eye at approximate 5 hour intervals QID during the non-sleep period for a duration of 12 weeks.
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Age, Continuous [Mean (Standard Deviation); unit: Years] | 76.3 (6.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 5
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Central Retinal Lesion Thickness (CRT) as Measured by Optical Coherence Tomography (OCT) at Day 29
Description: CRT was the distance between the inner limiting membrane of the retina and the inner border of the retinal pigment epithelium/choriocapillaris band, inclusive of sub retinal fluid, measured in the central 1 millimeter (mm) of the Cube scan. OCT assessments were performed using SPECTRALIS spectral domain OCT. Images were evaluated by investigator for safety monitoring, and by a central reading center for eligibility determination and pharmacodynamics (PD) effects. Observed case (OC) data set was used for analysis in this analysis dataset, a missing assessment at any scheduled time point was considered unevaluable, was not imputed and was not included in data analysis. Baseline was defined as the assessments performed between Day -3 to -1. Change from Baseline was calculated by subtracting the baseline value from the individual post-randomization value at Day 29.
Time Frame: Baseline (Week 0) and Day 29
Population: The Intent-to-treat (ITT) Population comprised of any participant who received at least one dose of study medication. Only those participants with data available at the indicated time point were analyzed. OC dataset was used for analysis.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 13
Microns | 37.91 (89.692)

2. Primary Outcome: Change From Baseline in Best Correct Visual Acuity (BCVA) as Measured by the Number of Letters Determined by Electronic Early Treatment Diabetic Retinopathy [ETDRS] Study Visual Acuity (EVA) at Day 29
Description: BCVA was measured in the study eye using the EVA chart starting at a test distance of 4 meters. The BCVA score is the number of letters read correctly by the participant. A decrease in the BCVA score indicates a worsening of vision while higher scores indicates improvement of VA. Baseline was defined as the assessments performed between Day -3 to -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization value at Day 29.
Time Frame: Baseline (Day -3 to -1) and Day 29
Population: ITT Population. Only those participants with data available at the indicated time point were analyzed. OC dataset was used for analysis.
Measure: Mean (Standard Deviation); unit: Count of letters
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 13
Count of letters | 0.07 (9.973)

3. Secondary Outcome: Change From Baseline in Central Retinal Lesion Thickness (CRLT) Over Time
Description: CRLT was the manual measurement of the distance between the inner limiting membrane of the retina and the inner border of the choriocapillaris, inclusive of subretinal or sub-retinal pigment epithelium fluid collections and of the thickness of any observable choroidal neovascular membrane or scar tissue, evaluated in the central 1 mm of the Cube scan. OCT assessments were performed using SPECTRALIS spectral domain OCT. Baseline was defined as the assessments performed between Day -3 to -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization value at Day 29.
Time Frame: Baseline (Week -3 to -1) Up to Follow-up (Day 102)
Population: ITT Population. Only those participants available at the specified time points were analyzed. OC dataset was used for analysis.
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Microns
  CRLT at Week 1 | -3.97 (93.420)
  CRLT at Week 2 | -6.39 (93.420)
  CRLT at Week 3: number analyzed (Participants) | 14
  CRLT at Week 3 | 15.15 (86.646)
  CRLT at Week 4: number analyzed (Participants) | 13
  CRLT at Week 4 | 31.72 (88.289)
  CRLT at Week 6: number analyzed (Participants) | 10
  CRLT at Week 6 | 51.22 (84.679)
  CRLT at Week 8: number analyzed (Participants) | 8
  CRLT at Week 8 | 15.48 (82.304)
  CRLT at Week 12: number analyzed (Participants) | 6
  CRLT at Week 12 | -1.57 (75.216)
  CRLT at Follow-up: number analyzed (Participants) | 11
  CRLT at Follow-up | -8.42 (91.346)

4. Secondary Outcome: Change From Baseline in Intraretinal (IR) or Subretinal (SR) Fluid Thickness, Intraretinal Cysts or Serous Retinal Pigment Epithelial Detachment (PED Thickness) Over Time
Description: OCT was used for the determination of retinal morphology changes in the study eye which included assessments of SR fluid (an exudate between the retina and choroid from various sources including the vitreous cavity, subarachnoid space, or abnormal vessels) and PED (retinal pigment epithelium separates from the underlying Bruch's membrane due to the presence of blood, serous exudate, drusen, or a neovascular membrane). Baseline was defined as the assessments performed between Day -3 to -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization value at Day 29.
Time Frame: Baseline (Week -3 to -1) Up to Follow-up (Day 102)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Microns
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Microns
  SR fluid thickness at Week 1: number analyzed (Participants) | 17
  SR fluid thickness at Week 1 | -34.79 (70.781)
  SR fluid thickness at Week 2: number analyzed (Participants) | 18
  SR fluid thickness at Week 2 | -29.32 (71.654)
  SR fluid thickness at Week 3: number analyzed (Participants) | 13
  SR fluid thickness at Week 3 | -0.22 (67.074)
  SR fluid thickness at Week 4: number analyzed (Participants) | 12
  SR fluid thickness at Week 4 | 5.69 (67.938)
  SR fluid thickness at Week 6: number analyzed (Participants) | 10
  SR fluid thickness at Week 6 | 28.05 (67.192)
  SR fluid thickness at Week 8: number analyzed (Participants) | 7
  SR fluid thickness at Week 8 | 35.25 (64.689)
  SR fluid thickness at Week 12: number analyzed (Participants) | 4
  SR fluid thickness at Week 12 | 1.72 (57.734)
  SR fluid thickness at Follow-up: number analyzed (Participants) | 8
  SR fluid thickness at Follow-up | 8.43 (70.329)
  PED thickness at Week 1: number analyzed (Participants) | 12
  PED thickness at Week 1 | 4.01 (56.669)
  PED thickness at Week 2: number analyzed (Participants) | 12
  PED thickness at Week 2 | 4.47 (56.669)
  PED thickness at Week 3: number analyzed (Participants) | 9
  PED thickness at Week 3 | 14.00 (53.040)
  PED thickness at Week 4: number analyzed (Participants) | 9
  PED thickness at Week 4 | 7.16 (54.843)
  PED thickness at Week 6: number analyzed (Participants) | 5
  PED thickness at Week 6 | 37.93 (49.035)
  PED thickness at Week 8: number analyzed (Participants) | 3
  PED thickness at Week 8 | 36.57 (46.786)
  PED thickness at Week 12: number analyzed (Participants) | 3
  PED thickness at Week 12 | -32.68 (46.509)
  PED thickness at Follow-up: number analyzed (Participants) | 7
  PED thickness at Follow-up | -19.04 (56.214)

5. Secondary Outcome: Change From Baseline in BCVA Over Time
Description: as for outcome 2
Time Frame: Baseline (Week -3 to -1) Up to Follow-up (Day 102)
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Letters
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Letters
  Week 1 | 0.26 (11.015)
  Week 2 | 0.26 (11.015)
  Week 3: number analyzed (Participants) | 14
  Week 3 | -1.47 (9.927)
  Week 4: number analyzed (Participants) | 13
  Week 4 | 0.07 (9.973)
  Week 6: number analyzed (Participants) | 10
  Week 6 | 1.76 (9.345)
  Week 8: number analyzed (Participants) | 8
  Week 8 | 0.63 (8.912)
  Week 12: number analyzed (Participants) | 6
  Week 12 | -0.85 (8.069)
  Follow-up: number analyzed (Participants) | 11
  Follow-up | -5.49 (10.388)

6. Secondary Outcome: Change From Baseline in the Area of Choroidal Neovascular (CNV) Size and CNV Total Lesion Complex Size as Measured by Fluorescein Angiography (FA) at Day 29
Description: CNV was the measurement of the combined classic and occult neovascular lesion including areas of classic neovascularization, late staining of undetermined origin and fibrovascular PED. CNV total lesion complex size was the measurement of the entire lesion including classic and occult neovascular components as well as contagious blood and/or blocked fluorescence and/or serous PED. FA uses fundus photography (FP) to capture images of injected dye circulating throughout the retinal blood vessels to assess leaking, swelling/circulation problems caused by various eye diseases like diabetic retinopathy and wet macular degeneration. A fluorescein angiogram was obtained at Day 29. Images were evaluated by investigator for eligibility and by a central reading center for determination of PD effect. Baseline was defined as the assessments performed between Day -3 to -1. Change from Baseline was calculated by subtracting the Baseline value from the individual post-randomization value at Day 29.
Time Frame: Baseline (Day -3 to -1) and Day 29
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: millimeter square
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 13
millimeter square
  CNV Size at Week 4 | 1.38 (2.902)
  CNV total lesion complex size at Week 4 | 1.37 (2.892)

7. Secondary Outcome: Number of Participants With Change in Charactertsics (Atrophy, Pigment, SR Hemorrhage, IR Hemorrhage, SR Fluid and Fibrosis) as Measured by FP
Description: Fundus photography involves capturing of images of the center of the very back inner wall of the eye - the retina, optic nerve, macula and main retinal blood vessels. The parameters assessment were heme SR hemorrhage (absence or presence at the location), heme IR hemorrhage (absence or presence at the location), SR fluid (absence or presence at location), fibrosis (absence or presence at location), atrophy (absence or presence of atrophic changes) and pigment (absence or presence at location). A protocol set of fundus photographs were obtained at Day 29. Images were read by the investigator for eligibility determination, and by a central reading center for determination of PD effect. Data has been presented for number of participants with changes in eye characteristics in the study eye at Day 29.
Time Frame: Day 29
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 13
Participants
  Atrophy at Week 4 | 0
  Pigment at Week 4 | 12
  Heme (SR) at Week 4 | 10
  Heme (IR) at Week 4 | 1
  SR fluid at Week 4 | 13
  Fibrosis at Week 4 | 1

8. Secondary Outcome: Number of Participants Who Received Rescue Medication
Description: At any time during the study, including the follow-up period, rescue treatment (standard of care) was given based on the clinical judgment of the investigator. Rescue treatment was to be strongly considered for participants whose center subfield thickness had increased by >50 microns from the lowest value on study or whose BCVA decreased by more than 5 letters compared to baseline and who also had persistent fluid by OCT. Data has been reported for the number of participants with their percentages who required any rescue medication administration until follow-up.
Time Frame: Up to follow-up (Day 102)
Population: Safety Population comprised of any participant who received at least one dose of study medication.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Participants | 9

9. Secondary Outcome: Number of Participants With Ocular Adverse Events (AEs), Non-ocular AEs, Serious Ocular AEs and Serious Non-ocular AEs
Description: An AE is defined as any untoward medical occurrence in a participant or clinical investigation participant, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding), symptom, or disease (new or exacerbated) temporally associated with the use of a medicinal product. An SAE is defined as any untoward medical occurrence that, at any dose, results in death, is life threatening, requires hospitalization or prolongation of existing hospitalization, results in disability/incapacity, is a congenital anomaly/birth defect, may jeopardize the participant or require medical or surgical intervention to prevent one of the other outcomes listed in the definition above, or is an event of possible drug-induced liver injury.
Time Frame: Until Follow-up (Day 102)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Participants
  Any Ocular AE | 8
  Any Ocular SAE | 0
  Any Non-Ocular AE | 9
  Any Non-Ocular SAE | 0

10. Secondary Outcome: Number of Participants With Values of Potential Clinical Concern for Ocular Assessments on General Ophthalmic Examination
Description: A complete eye examination was performed to include the following: Examination of eyelids and lashes (including meibomian glands), Pupil, motility and confrontation visual field examination, Slit lamp evaluation of anterior ocular structures (including conjunctiva, tear film, cornea with fluorescein staining, anterior chamber, iris, lens, and anterior vitreous), Intraocular pressure (IOP) measurement and Dilated Fundus Examination (Indirect ophthalmoscopy and slit lamp biomicroscopy). Data has been presented in a consolidated format for the total number of participants with values of potential clinical concern for complete ophthalmic examinations until Day 102.
Time Frame: Up to Follow-up (Day 102)
Population: Safety Population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Participants | 0

11. Secondary Outcome: Number of Participants With Vital Sign Data of Potential Clinical Concern
Description: Vital sign assessments included systolic blood pressure, diastolic blood pressure and heart rate. The potential clinical concern range for systolic blood pressure was <85 and >160 millimeters of mercury, diastolic blood pressure <45 and > 100 millimeters of mercury, heart rate <40 and >110 beats per minute. Data has been presented in a consolidated format for the total number of participants with values of potential clinical concern for systolic blood pressure, diastolic blood pressure and heart rate until Day 102.
Time Frame: Up to Follow-up (Day 102)
Population: Safety Population
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Participants
  Systolic blood pressure | 2
  Diastolic blood pressure | 0
  Heart rate | 0

12. Secondary Outcome: Number of Participants With Clinical Chemistry and Hematology Data of Potential Clinical Concern
Description: Clinical chemistry parameters included albumin, alkaline phosphatase, alanine amino transferase, aspartate amino transferase, direct bilirubin, total bilirubin, calcium, chloride, carbon dioxide, creatinine, thyroxine (T3 free), gamma glutamyl transferase, glucose, potassium, sodium, total protein, total T3, urea, uric acid while hematology included basophils, eosinophils, hemoglobin, hematocrit, lymphocytes, mean corpuscle hemoglobin concentration, mean corpuscle hemoglobin, mean corpuscle volume, monocytes, segmented neutrophils, total neutrophils, platelet count, red blood cell count, reticulocytes and white blood cell count. The potential clinical concern ranges were as follows: glucose-low <3 and high >9 millimoles per liter (mmol/L), carbon dioxide-low <18 and high >34 mmol/L, lymphocyte-low <0.8 giga per liter (G/L) and platelet count was <100 and high >550 G/L. Data has been presented for the number of participants with values high and low of potential clinical concern.
Time Frame: Up to Follow-up (Day 102)
Population: Safety population.
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Participants
  Glucose high | 1
  Carbon dioxide low | 2
  Lymphocyte low | 1
  Platelet count low | 1

13. Secondary Outcome: Number of Participants With Abnormal Urinalysis Data by Urine Microscopy and Dipstick Analysis
Description: Urinalysis measurements included assessments for red blood cells and white blood cells via microscopic examination while assessments for urine protein by standard dipstick analysis. Data has been presented for the number of participants with abnormal urinalysis results.
Time Frame: Up to Follow-up (Day 102)
Population: Safety Population. Only those participants available at the specified time points were analyzed,
Measure: Count of Participants; unit: Participants
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
Participants
  Red blood cells 3-5 at Week 2: number analyzed (Participants) | 1
  Red blood cells 3-5 at Week 2 | 1
  Red blood cells 0-1 at Week 4: number analyzed (Participants) | 3
  Red blood cells 0-1 at Week 4 | 1
  Red blood cells 1-3 at Week 4: number analyzed (Participants) | 3
  Red blood cells 1-3 at Week 4 | 1
  Red blood cells 25-50 at Week 4: number analyzed (Participants) | 3
  Red blood cells 25-50 at Week 4 | 1
  Red blood cells 1-3 at Follow-up: number analyzed (Participants) | 5
  Red blood cells 1-3 at Follow-up | 1
  Red blood cells 5-10 at Follow-up: number analyzed (Participants) | 5
  Red blood cells 5-10 at Follow-up | 2
  White blood cells 3-5 at Week 2: number analyzed (Participants) | 1
  White blood cells 3-5 at Week 2 | 1
  White blood cells 1-3 at Week 4: number analyzed (Participants) | 3
  White blood cells 1-3 at Week 4 | 1
  White blood cells 5-10 at Week 4: number analyzed (Participants) | 3
  White blood cells 5-10 at Week 4 | 1
  White blood cells 10-15 at Follow-up: number analyzed (Participants) | 5
  White blood cells 10-15 at Follow-up | 1
  White blood cells 50-100 at Follow-up: number analyzed (Participants) | 5
  White blood cells 50-100 at Follow-up | 1
  Urine protein 2+ at Week 4: number analyzed (Participants) | 13
  Urine protein 2+ at Week 4 | 1
  Urine protein 1+ at Week 12: number analyzed (Participants) | 6
  Urine protein 1+ at Week 12 | 1
  Urine protein 2+ at Week 12: number analyzed (Participants) | 6
  Urine protein 2+ at Week 12 | 1
  Urine protein 1+ at Follow-up: number analyzed (Participants) | 17
  Urine protein 1+ at Follow-up | 1
  Urine protein 3+ at Follow-up: number analyzed (Participants) | 17
  Urine protein 3+ at Follow-up | 1

14. Secondary Outcome: Summary of Plasma Pazonib Concentration
Description: Throughout the study, 1 to 4 blood samples (2 mL) were collected from each participants for the analysis of plasma pazopanib concentrations between 0.55 to 10.83 hours post-dose on Weeks 2, 3, 4, 6 (unplanned), 8 (unplanned) and 12. The concentrations from the three blood samples per participant were averaged and then the values were averaged through all the participants. Blood samples were collected without restriction for the time interval between blood draw and the last dose of pazopanib eye drops.
Time Frame: Up to Week 12
Population: Pharmacokinetic Population was defined as participants in the ITT Population for whom a pharmacokinetic sample was obtained and analyzed. Only those participants available at the specified time points were analyzed.
Measure: Mean (Standard Deviation); unit: nanograms per milliliter
Arm/Group | Pazopanib 10 mg/mL QID
Number analyzed (Participants) | 19
nanograms per milliliter
  Week 2 | 279.0 (171.66)
  Week 3: number analyzed (Participants) | 7
  Week 3 | 323.9 (216.77)
  Week 4: number analyzed (Participants) | 14
  Week 4 | 360.5 (215.80)
  Week 6: number analyzed (Participants) | 1
  Week 6 | 498.0 (NA) — Standard could was not computed as a single participant was analyzed.
  Week 8: number analyzed (Participants) | 1
  Week 8 | 150.0 (NA) — Standard could was not computed as a single participant was analyzed.
  Week 12: number analyzed (Participants) | 6
  Week 12 | 255.3 (170.06)

ADVERSE EVENTS:
Time Frame: Up to Follow-up (Day 102)
Description: Safety population was used for analysis.
Arm/Group | Pazopanib 10 mg/mL QID
All-Cause Mortality (participants affected / at risk) | 0/19
Serious Adverse Events (participants affected / at risk) | 0/19
Other Adverse Events (participants affected / at risk) | 17/19
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pazopanib 10 mg/mL QID (N=19)
Age-related macular degeneration (Eye disorders) | 2
Macular oedema (Eye disorders) | 1
Ocular Hypertension (Eye disorders) | 1
Retinal haemorrhage (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Instillation site pain (General disorders) | 3
Nausea (Gastrointestinal disorders) | 1
Oesophageal obstruction (Gastrointestinal disorders) | 1
Tooth infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Skeletal injury (Injury, poisoning and procedural complications) | 1
Platelet count decreased (Investigations) | 1
Protein urine present (Investigations) | 1
Red blood cells urine positive (Investigations) | 1
Urine protein/creatinine ratio increased (Investigations) | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Tendonitis (Musculoskeletal and connective tissue disorders) | 1
Torticollis (Musculoskeletal and connective tissue disorders) | 1
Depression (Psychiatric disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyshponia (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.